CLINICAL TRIAL: NCT05444283
Title: Large Scale Genome Sequencing and Integrative Analyses to Define Genomic Predictors of Recurrent Pregnancy Loss
Brief Title: Genomic Predictors of Recurrent Pregnancy Loss
Acronym: GPRPL
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Johns Hopkins University (Other); University of Texas at Austin (Other); Penn State University (Other); Northwestern University (Other); The University of Texas Health Science Center at San Antonio (Other); Wayne State University (Other); Columbia University (Other); University of Colorado, Denver (Other); University of Chicago (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 2000029802; 1R01HD105267-01 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Products of conception and blood or saliva of one or both biological parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goals of this proposal are to determine the genetic architecture of recurrent pregnancy loss (RPL) and to discover genomic predictors of RPL.

DETAILED DESCRIPTION:
The following specific aims are proposed:

Aim 1: Collect clinically well-characterized samples from two distinct cohorts of participants with unexplained recurrent pregnancy loss (RPL).

* Cohort A will consist of trios (product of conception (POC), biological mother, and biological father) with unexplained RPL. Specifically, a cohort of up to 500 rigorously phenotyped trios will be recruited, for which couples' RPL is not attributable to known causes. POC tissues and parental DNA samples (blood or saliva) will be collected. If necessary for the purpose of determining the pathogenicity of sequence variants identified in the trio, collecting DNA samples from other family members after consent will also be considered. The study team may also request DNA or POC tissues from prior pregnancy loss(es) if available.
* Cohort B will consist of up to 100 women with a history of three or more pregnancy losses, with or without a liveborn child, and no known etiology. For these participants, DNA samples (blood or saliva) will be collected from the mothers. If high-impact variants are identified, DNA samples from parents or siblings may be collected for segregation analysis after consent.

Aim 2: Whole genome sequencing (WGS) will be performed at the Yale Center for Genome Analysis (YCGA), along with bioinformatic analyses to identify pathogenic variants in both cohorts. For Cohort A, analyses will focus on pathogenic variants identified in RPL trios, and for Cohort B, analyses will focus on variants associated with maternal effect genes in the mothers. Pathogenic variants will be comprehensively defined, and fully annotated variant maps will be generated for all included samples to provide the substrate for subsequent novel gene discovery and, ultimately, the development of clinical diagnostic tests.

ELIGIBILITY:
Cohort A - Fetal Intolerome Cohort

Inclusion Criteria:

* Women with loss of a current singleton pregnancy at < 20 0/7 weeks gestation, documented by ultrasonography or histopathological examination
* History of one or more prior pregnancy losses
* Euploid current pregnancy confirmed by karyotype, microarray, or STORK (Short-read Transpore Rapid Karyotyping) sequencing Note: A limited number of aneuploid losses will be included as part of the pilot phase

Exclusion Criteria:

* History of parental karyotype abnormalities
* History of antiphospholipid antibody syndrome
* Evidence of uncontrolled diabetes
* Evidence of uncontrolled thyroid disease
* History of autoimmune disease related to pregnancy loss (e.g., systemic lupus erythematosus, rheumatoid arthritis)
* History of uterine anomalies
* History of cervical insufficiency

Cohort B - Maternal Effect Gene Cohort

Inclusion Criteria:

- Women with a history of three or more pregnancy losses of unknown cause, with or without a liveborn child

Exclusion Criteria:

- Known etiology for pregnancy loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples who have had two or more previous pregnancy losses and have undiagnosed cause of recurrent pregnancy loss.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine genetic etiology for Recurrent Pregnancy Loss | 5 years
  The WGS tool will be used to analyze the POC sample and parental blood samples to determine the clinical reportable genetic cause for RPL

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Gaelle Massoud, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - University of Texas at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No